CLINICAL TRIAL: NCT05663489
Title: Neurobiological Markers of Treatment Response for Anxiety and OCD
Status: Recruiting | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Oslo (Other); Amsterdam UMC, location VUmc (Other); University of North Carolina, Chapel Hill (Other); Harvard Medical School (HMS and HSDM) (Other); University of Bergen (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BCBP-1
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Obsessive-Compulsive Disorder; Social Anxiety Disorder; Panic Disorder
Keywords: MRI; epigenetics; genetics
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Phobia, Social; Panic Disorder | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with obsessive-compulsive, social anxiety or panic disorder: Patients with obsessive-compulsive disorder. The MRI substudy will also include patients with social anxiety or panic disorder
  Interventions: Behavioral: Bergen 4-Day Treatment (B4DT)
- For MRI substudy: Healthy controls: Healthy controls demographically matched to the patient group on age, sex and years of education

INTERVENTIONS:
Behavioral: Bergen 4-Day Treatment (B4DT) — A concentrated and exposure-based psychological treatment over four consecutive days
  Groups: Patients with obsessive-compulsive, social anxiety or panic disorder

SUMMARY:
Obsessive-compulsive disorder (OCD) and anxiety disorders are common and debilitating conditions which are often chronic when treatment is not provided. International guidelines recommend cognitive behavioral therapy (CBT) as the first-line treatment, and research has shown that CBT can be delivered over a concentrated period of time. The Bergen 4-Day Treatment (B4DT) is an exposure-based treatment which is delivered over four consecutive days. B4DT has been shown to induce rapid and long-lasting remission in around 70% of patients. This provides a platform for studying psychological and neurobiological changes associated with treatment response and non-response. The present study will investigate longitudinal changes in psychological measures and DNA methylation in patients who receive the B4DT, as well as a subset will also undergo multimodal brain imaging.

DETAILED DESCRIPTION:
The primary study will include 500 OCD patients who will receive the B4DT. Symptom severity will be prospectively measured before treatment, approximately 10 days after treatment and three months after treatment. Saliva samples will be collected for later extraction of DNA methylation during the first day of treatment, the last day of treatment, and three months after treatment. A substudy will use multimodal magnetic resonance imaging (MRI) before treatment, approximately 10 days after treatment and three months after treatment. The substudy will also 100 patients with social anxiety disorder or panic disorder for DNA methylation and MRI, as well as 50 healthy controls for MRI. Clinical data will be collected from a consent-based quality register ("Kvalitetsregister for konsentrerte behandlingsformat").

The aim of the study is to investigate changes in DNA methylation as well as functional and structural brain networks that occur in patients undergoing B4DT, and to correlate these changes with immediate and long-term response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with obsessive-compulsive disorder, panic disorder or social anxiety disorder using DSM-5 criteria
* Referred to National Clinic for 4-Day Treatment, Haukeland University Hospital, Bergen, Norway
* Consented to participate in the "Kvalitetsregister for konsentrerte behandlingsformat"

Exclusion Criteria:

* Suicidal, ongoing mania, primary eating disorder, intellectual disability, ongoing psychosis, ongoing substance abuse

For MRI substudy:

Inclusion Criteria:

- For the healthy controls, no previous or current psychiatric disorders as detected by the Mini International Neuropsychiatric Interview (MINI)

Exclusion Criteria:

- MRI incompatibility (e.g. pregnancy, metal implants)

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study includes patients with OCD, panic disorder or social anxiety disorder which will receive the Bergen 4-Day Treatment (B4DT) in Norway. Healthy controls are also recruited for the MRI substudy
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-03-23 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2027-12-11 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | Before treatment
  Symptom severity of obsessive-compulsive disorder
Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | approximately 10 days after treatment
  Symptom severity of obsessive-compulsive disorder
Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | three months after treatment
  Symptom severity of obsessive-compulsive disorder
Panic Disorder Severity Scale (PDSS) | Before treatment
  Symptom severity of panic disorder
Panic Disorder Severity Scale (PDSS) | approximately 10 days after treatment
  Symptom severity of panic disorder
Panic Disorder Severity Scale (PDSS) | three months after treatment
  Symptom severity of panic disorder
Liebowitz Social Anxiety Scale (LSAS) | Before treatment
  Symptom severity of social anxiety disorder
Liebowitz Social Anxiety Scale (LSAS) | approximately 10 days after treatment
  Symptom severity of social anxiety disorder
Liebowitz Social Anxiety Scale (LSAS) | three months after treatment
  Symptom severity of social anxiety disorder

SECONDARY OUTCOMES:
DNA Methylation | Before treatment
  Samples of saliva will be collected for genome-wide methylation and profiling will be carried out using the Illumina Infinium MethylationEPIC BeadChip system
DNA Methylation | approximately 10 days after treatment
  Samples of saliva will be collected for genome-wide methylation and profiling will be carried out using the Illumina Infinium MethylationEPIC BeadChip system
DNA Methylation | three months after treatment
  Samples of saliva will be collected for genome-wide methylation and profiling will be carried out using the Illumina Infinium MethylationEPIC BeadChip system
Magnetic Resonance Imaging | Before treatment
  Brain functional and structural MRI will be collected for a subset of 100 OCD and 100 anxiety disorder patients as well as 50 healthy controls
Magnetic Resonance Imaging | approximately 10 days after treatment
  Brain functional and structural MRI will be collected for a subset of 100 OCD and 100 anxiety disorder patients as well as 50 healthy controls
Magnetic Resonance Imaging | three months after treatment
  Brain functional and structural MRI will be collected for a subset of 100 OCD and 100 anxiety disorder patients as well as 50 healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Bjarne Hansen, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Bergen Center for Brain Plasticity, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: No